CLINICAL TRIAL: NCT06413589
Title: Efficacy of SMOF Lipid in the Management of Acute Poisoning With Clozapine Secondary IDs:
Brief Title: Efficacy of SMOF Lipid in the Management of Acute Poisoning With Clozapine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMOF in clozapine toxicity
Record Dates: First submitted 2024-04-18; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Acute Poisoning
Keywords: clozapine poisoning; SMOF lipid; lipophilic agents

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): The first group constitutes the control group that was administered the standard treatment protocol for clozapine toxicity.
  Interventions: Other: standard treatment for clozapine toxicity
- SMOF lipid treated group (Active Comparator): The second group received the SMOF lipid infusion in addition to the standard protocol.Drug: SMOF lipid 20% SMOF 20%; a blend of soybean oil, medium-chain triglycerides, olive oil, and fish oil, is a new lipid emulsion product that was provided as a bolus dose of 1.5ml/kg for one hour, followed by a maintenance dose of 6 ml/kg for a period of four hours to the active comparator group
  Interventions: Other: SMOF lipid 20%

INTERVENTIONS:
Other: SMOF lipid 20% — Drug: SMOF lipid 20% SMOF 20%, a blend of soybean oil, medium-chain triglycerides, olive oil, and fish oil, is a new lipid emulsion product that was provided as a bolus dose of 1.5ml/kg for one hour, followed by a maintenance dose of 6 ml/kg for a period of four hours to the active comparator group
  Arms: SMOF lipid treated group
Other: standard treatment for clozapine toxicity — Hypotension was initially treated with isotonic crystalloid; vasopressors were utilised if intravenous fluids failed to restore the hypotension. This was in the form of norepinephrine with a dose of 0.05 μg/kg/min and titrated till reaching the goal mean arterial pressure (>65 mmHg) [29].
  Those experiencing seizures due to CBZ overdose were treated with benzodiazepines (diazepam) at a dose of 10-20 mg. Benzodiazepines are considered allosteric modulators of the gamma-aminobutyric acid channel.
  MDAC (50 grammes every six hours) was given to all patients in the current study. Those with severe poisoning were given the MDAC after securing the airway with a cuffed endotracheal tube
  Arms: control group

SUMMARY:
The goal of the current study was to evaluate whether SMOF lipid administration could be used as an adjuvant therapy to treat acute, moderate-to-severe clozapine poisoning.

DETAILED DESCRIPTION:
Antipsychotics, a class of drugs primarily used to treat schizophrenia and various mood disorders, including bipolar disorder, encompass a medication like clozapine. Clozapine stands out among antipsychotics due to its lower incidence of extrapyramidal symptoms, such as tardive dyskinesia, and its effectiveness in addressing negative symptoms of schizophrenia.

Recent data from the American Association of Poison Control Centers (AAPCC) highlight sedatives/hypnotics/antipsychotics as among the top five frequently encountered xenobiotics in human exposure cases. This class of drugs has seen a notable uptick in incidence over the past 18 years. In Egypt, studies from institutions like Tanta University Poison Control Centre (TUPCC) and the National Poisoning Center in Cairo have identified acute clozapine poisoning as a common occurrence within cases of pharmaceutical drug poisonings affecting the central nervous system.

Clozapine toxicity manifests across multiple organ systems, with the central nervous system (CNS) and cardiovascular system (CVS) being most significantly impacted. Common symptoms include pronounced sedation, confusion, delirium, tachycardia, and mild hypotension.

Because there is no definitive antidote for clozapine poisoning, poison control centres recommend supportive therapy based on the patient's clinical condition and multiple-dose activated charcoal (MDAC) as a specific intervention for enhanced elimination. Nevertheless, the elimination of the drug from the body can be prolonged.

The scarcity of physiological antidotes for acute poisonings encourages toxicologists to supplement standard supportive treatment protocols with promising agents that tend to improve morbidity and mortality.

In this context, intravenous lipid emulsions (ILE) are mainly used as a source of energy and essential fatty acids in patients requiring parenteral nutrition. Apart from their nutritional value, lipid emulsion therapy is becoming increasingly popular in critical care settings as a treatment for toxicity with lipophilic agents, particularly when the standard remedies are ineffective.

Following the encouraging outcomes of using ILEs for the treatment of local anaesthetic systemic toxicity, subsequent studies reported the therapeutic effect of ILEs in acute poisonings with other xenobiotics. However, the evidence for the potential effectiveness of ILE in clinical toxicology consists mainly of case reports and experimental studies.

ILE may be suitable for the treatment of clozapine toxicity due to its lipid solubility.

SMOF 20%, a blend of soybean oil, medium-chain triglycerides, olive oil, and fish oil, is a new lipid emulsion product that has shown better therapeutic results regarding parentral nutrition when compared with traditional ones such as Intralipid® 20%. It has been associated with decreased oxidative injury, improved liver function, and increased antioxidant activity

ELIGIBILITY:
Inclusion Criteria:

The patients were enrolled in the study in accordance with the following:

Gender and age: adult symptomatic males and females. Patients were admitted within 12 hours of exposure to the poison. Patients received no prior treatment before admission. Patients with moderate-to-severe carbamazepine poisoning according to the Poisoning Severity Score (PSS) Patients classified as high-risk (HR) with anti-depressant overdose risk assessment (ADORA) criteria.

Exclusion Criteria:

Patients were excluded if they had any of the following conditions:

pregnant and lactating women. Patients with major medical conditions (e.g. diabetes mellitus), cardiovascular disease, renal, or hepatic failure).

Patients suffering from hyperlipidemia. Malignancy. Co-ingestion.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Improvement in Conscious Levels Measured by Glasgow Coma Scale (GCS) | participants were monitored within 24 hours from admission to the hospital
  This study evaluates the efficacy of SMOF lipid 20% in improving conscious levels among participants with acute clozapine poisoning within 24 hours. Conscious level improvement is assessed using the Glasgow Coma Scale (GCS), a widely recognised tool for neurological assessment. The GCS measures eye opening, verbal response, and motor response. The minimum value is 3 and the maximum value is 15, with higher scores indicating better conscious levels. The study aims to determine the extent of improvement in GCS scores following SMOF lipid administration, providing valuable insights into its effectiveness in enhancing neurological function.
Assessment of Intubation Requirement Using APACHE | participants were assessed within 24 hours from admission to the hospital
  This study investigates the requirement for intubation and mechanical ventilation among participants with acute clozapine poisoning using multiple clinical assessment tools, including the Glasgow Coma Scale (GCS) and Acute Physiology and Chronic Health Evaluation (APACHE). The GCS evaluates the level of consciousness based on eye opening, verbal response, and motor response, with lower scores indicating a higher likelihood of intubation and mechanical ventilation. The APACHE score assesses the severity of illness and predicts the need for respiratory support, with higher scores indicating an increased risk of respiratory failure and the requirement for intervention.
Length of Intensive Care Unit (ICU) Stay | up to one month
  This study evaluates the length of stay in the Intensive Care Unit (ICU) among participants with acute clozapine poisoning. The length of the ICU stay is defined as the duration from the time of admission to the ICU to discharge from the ICU in days. Participants will be monitored throughout their hospitalisation period, and the length of their ICU stay will be recorded. The study aims to assess the impact of SMOF lipid administration on the duration of ICU stays, providing insights into its effectiveness in optimising resource utilisation and patient management. Understanding the factors influencing the length of the ICU stay may contribute to improved healthcare delivery and patient outcomes in acute clozapine poisoning.
length of hospital stay | up to one month
  This study evaluates the length of stay in the hospital among participants with acute clozapine poisoning. The length of stay is defined as the duration from the time of admission to the hospital to discharge from the hospital in days. Participants will be monitored throughout their hospitalisation period, and the length of their hospital stay will be recorded. The study aims to assess the impact of SMOF lipid administration on the duration of hospital stays, providing insights into its effectiveness in optimising resource utilisation and patient management. Understanding the factors influencing length of stay may contribute to improved healthcare delivery and patient outcomes in acute clozapine poisoning.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Sheta, professor, Study Chair — Alexandria University
Locations (1):
- Faculty of Medicine, Alexandria, Egypt

REFERENCES:
- [Background] Jaffal K, Chevillard L, Megarbane B. Lipid Emulsion to Treat Acute Poisonings: Mechanisms of Action, Indications, and Controversies. Pharmaceutics. 2023 May 3;15(5):1396. doi: 10.3390/pharmaceutics15051396. PMID 37242638
- [Background] Elgazzar FM, Elgohary MS, Basiouny SM, Lashin HI. Intravenous lipid emulsion as an adjuvant therapy of acute clozapine poisoning. Hum Exp Toxicol. 2021 Jul;40(7):1053-1063. doi: 10.1177/0960327120983873. Epub 2021 Jan 5. PMID 33401984
- [Background] Taftachi F, Sanaei-Zadeh H, Sepehrian B, Zamani N. Lipid emulsion improves Glasgow coma scale and decreases blood glucose level in the setting of acute non-local anesthetic drug poisoning--a randomized controlled trial. Eur Rev Med Pharmacol Sci. 2012 Mar;16 Suppl 1:38-42. PMID 22582483
- [Background] Ok SH, Sohn JT. Effect of lipid emulsion on acute clozapine poisoning-induced QT prolongation. Hum Exp Toxicol. 2021 Dec;40(12):2237-2239. doi: 10.1177/09603271211025598. Epub 2021 Jun 17. No abstract available. PMID 34137281